CLINICAL TRIAL: NCT02395523
Title: A Phase II Study Using Hypofractionated Proton Beam Radiotherapy for Inoperable Hepatocellular Carcinoma
Brief Title: Hypofractionated Proton Beam Radiotherapy for Inoperable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-15-042
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Proton Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Beam Therapy (Experimental): Definition of target volume:
  * Gross tumor volume (GTV) = gross tumor defined using a treatment planning CT scan
  * Clinical target volume (CTV) = GTV + internal target volume
  * Planning target volume (PTV) = CTV + 5 - 7 mm of lateral, craniocaudal, and anteroposterior margins.
  Radiation dose and planning
  * Prescription dose to PTV: 70 GyE /10 fx, 7GyE fraction dose, 5 days/week
  * Dose prescription : 95% isodose volume of prescribed dose encompassed PTV
  Interventions: Radiation: Proton Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — Definition of target volume:
  * Gross tumor volume (GTV) = gross tumor defined using a treatment planning CT scan
  * Clinical target volume (CTV) = GTV + internal target volume
  * Planning target volume (PTV) = CTV + 5 - 7 mm of lateral, craniocaudal, and anteroposterior margins.
  Radiation dose and planning
  * Prescription dose to PTV: 70 GyE /10 fx, 7GyE fraction dose, 5 days/week
  * Dose prescription : 95% isodose volume of prescribed dose encompassed PTV
  Other Names: Radiotherapy

SUMMARY:
This phase II study is to evaluate the effectiveness of hypofractionated proton beam therapy (PBT) for Hepatocellular Carcinoma patients in hepatitis B endemic area.

DETAILED DESCRIPTION:
The primary endpoint is local progression free survival. The trial is a single arm phase II trial with the historical arm. The expected 3-year local progression free survival for patient with HCC patients treated with proton beam therapy would be 80%. With a power of 80% and a type I error level of 10%, evaluable 40 patients are required to reject that the null hypothesis that true 3-year local progression free survival rate is ≤65%. Considering the 10% unevaluable patients due to loss of follow up, a total 45 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular Carcinoma diagnosed as (i) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level greater than 200 IU/ml and a radiologically compatible feature with HCC in one or more CT/MRI/angiograms, or (ii) the presence of risk factors including hepatitis B or C virus and liver cirrhosis, a serum a-fetoprotein (AFP) level less than 200 IU/ml, and a radiologically compatible feature with HCC in two or more CT/MRI/angiograms or (iii) histological confirmation
* Inoperable HCC or refusal to surgery
* Recurrent/residual tumor after other local treatments (local ablation therapy, or transarterial chemoemobolization, etc), or unsuitable/refusal to other treatments.
* Patients without evidence of extrahepatic metastasis
* The largest diameter of tumor should be less than 7cm, and the number of tumor ≤2
* The targeted tumors is more than 2cm away from the alimentary tract (i.e., stomach, duodenum, esophagus, small and large bowel)
* No previous treatment to target tumors by other forms of RT
* Liver function of Child-Pugh class A or B7 (Child-Pugh score of ≤7)
* Age of ≥18 years
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) score
* Required Entry Laboratory Parameters WBC count ≥ 1,500/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 30,000/mm3; and adequate hepatic function (total bilirubin ≤ 3.0 mg/dL; AST and ALT < 5.0× upper limit of normal; no uncontrolled ascites
* No serious comorbidities other than liver cirrhosis
* Signed informed consent form prior to study entry

Exclusion Criteria:

* There is evidence of extrahepatic metastasis.
* Age of <18 years
* Liver function of Child-Pugh class B8-9 and C (Child-Pugh score of >7)
* Previous history of other forms of RT adjacent to target tumors
* Poor performance status of 2 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* Multicentric HCCs, except for those with the following two conditions: (i) multinodular aggregating HCC that could be encompassed by single clinical target volume and within single clinical target volume; (ii) lesions other than targeted tumor that were judged as controlled with prior surgery and/or local ablation therapy.
* Pregnant or breast feeding status
* Previous history uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
local progression - free survival | Up to 5 year
  During PBT, patients were assessed weekly and after comletion of PBT at the 1st month, every 3months for the first 2years, every 6 months up to 5years. the tumor responses were assessed according to the modified response evaluation criteria in solid tumors criteria by comparing pre- and posst-PBT CT/MRI scans, and the severity of adverse deffects was graded using the common terminology criteria for adverse events(ver 4.0)

SECONDARY OUTCOMES:
overall survival | Up to5 years until study closed
  During PBT, patients were assessed weekly and after com;letion of PBT at the 1st month, every 3months for the first 2years, every 6 months up to 5years. the tumor responses were assessed according to the modified response evaluation criteria in solid tumors criteria by comparing pre- and posst-PBT CT/MRI scans, and the severity of adverse deffects was graded using the common terminology criteria for adverse events(ver 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hyun Kim, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea